CLINICAL TRIAL: NCT06364371
Title: A Study of the Clinical Value of Dynamic Multi-omics Integration Model to Predict Neoadjuvant Therapy Response in Locally Advanced Rectal Cancer (T3-4NxM0)
Brief Title: Dynamic Multi-omics Integration Model to Predict Neoadjuvant Therapy Response in Locally Advanced Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: E2023210
Record Dates: First submitted 2024-04-02; First posted 2024-04-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Predictive Cancer Model; Pathologic Complete Response
Keywords: Magnetic resonance imaging; ctDNA; Histopathology slide; CEA
MeSH Terms: conditions — Pathologic Complete Response | interventions — Independent Medical Evaluation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: Patients with locally advanced (T3-4NxM0) rectal adenocarcinoma
  Interventions: Other: Medical examination

INTERVENTIONS:
Other: Medical examination — Eligible patients will be prospectively enrolled, and images of their pre-neoadjuvant treatment, during-treatment, and post-treatment preoperative magnetic resonance imaging (MRI) scans, histopathology slides stained with hematoxylin and eosin (H&E), carcinoembryonic antigen (CEA), and circulating tumor DNA (ctDNA) will be collected and annotated.

SUMMARY:
The goal of this observational study is to establish a dynamic multi-omics integration model for predicting pathological complete response (pCR) after neoadjuvant treatment in locally advanced (T3-4NxM0) rectal cancer, providing support for subsequent patient selection for the watch-and-wait strategy. The main question it aims to answer is:

What is the predictive value of this model to assess individual achievement of pathological complete response (pCR) after neoadjuvant treatment? Eligible patients will be prospectively enrolled, and the clinical features of their pre-neoadjuvant treatment, during-treatment, and post-treatment preoperative will be collected and annotated.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational phase II clinical study aimed at validating a dynamic multi-omics (imaging, pathology, molecular biomarkers) integration model for predicting pathological complete response (pCR) after neoadjuvant treatment in locally advanced (T3-4NxM0) rectal cancer. Specifically, the study aims to validate the predictive accuracy of the dynamic multi-omics prediction model and determine whether it outperforms other conventional prediction models based on single-modality imaging, pathology, and molecular biomarkers.

Eligible patients will be prospectively enrolled, and images of their pre-neoadjuvant treatment, during-treatment, and post-treatment preoperative magnetic resonance imaging (MRI) scans, histopathology slides stained with hematoxylin and eosin (H&E), carcinoembryonic antigen (CEA), and circulating tumor DNA (ctDNA) will be collected and annotated. MRI, H&E images, CEA, ctDNA, and their change features will be applied to the prediction model to assess individual achievement of pathological complete response (pCR) after neoadjuvant treatment. The predictive results will be further compared with the pathological tumor response obtained from resected specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed rectal adenocarcinoma;
2. Clinical stage T3-4NxM0, with or without positive Mesorectum Fascia(MRF), and with or without positive Extra-Mural Venous Invasion(EMVI);
3. Preoperative staging method: All patients undergo preoperative staging with enhanced CT. Criteria for mesorectal lymph node metastasis: Short axis ≥ 10mm lymph nodes or lymph node morphology and CT characteristics consistent with typical lymph node metastasis. Preoperative chest, abdominal CT, and pelvic MRI exclude distant metastases;
4. Absence of signs of intestinal obstruction; or relief of obstruction after proximal colon diversion surgery;
5. No history of previous colorectal surgery;
6. No history of previous chemotherapy or radiotherapy;
7. No history of previous biological therapy (such as monoclonal antibodies), immunotherapy [such as anti-programmed cell death protein 1(PD-1) antibodies, anti-PD-L1 antibodies, anti-PD-L2 antibodies, or anti-Cytotoxic T Lymphocyte-Associated Antigen-4(CTLA-4)], or other investigational drug therapy;
8. No history of previous hormonal therapy: no restrictions;
9. Signed informed consent form.

Exclusion Criteria:

1. Patients requiring antiarrhythmic therapy (excluding β-blockers or digoxin), symptomatic coronary artery disease, recent myocardial infarction within the past 6 months, or congestive heart failure exceeding New York Heart Association(NYHA) class II;
2. Poorly controlled severe hypertension;
3. History of HIV infection or active chronic hepatitis B or C (high viral DNA load);
4. Active pulmonary tuberculosis (TB) or receiving anti-TB treatment, or having received anti-TB treatment within the past year;
5. Other active clinically severe infections ;
6. Evidence of distant metastases outside the pelvis preoperatively;
7. Cachexia, organ decompensation;
8. History of pelvic or abdominal radiotherapy;
9. Multifocal colorectal cancer;
10. Patients requiring management for epileptic seizures (e.g., with steroids or antiepileptic therapy);
11. History of other malignant tumors within the past 5 years, excluding cured carcinoma in situ of the cervix or basal cell carcinoma of the skin;
12. Substance abuse or medical, psychological, or social conditions that may interfere with patient participation in the study or assessment of study results;
13. Presence of any active autoimmune disease or history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo or childhood asthma that has completely resolved and does not require any intervention in adulthood may be included; patients with asthma requiring bronchodilators for medical intervention cannot be included);
14. Vaccination with any anti-infective vaccine (e.g., influenza vaccine, varicella vaccine, etc.) within 4 weeks before enrollment;
15. Complications requiring long-term use of immunosuppressive drugs or systemic or local administration of corticosteroids with immunosuppressive effects (dose > 10mg/day of prednisone or equivalent corticosteroids);
16. Known or suspected allergy to the investigational drug or any medication administered related to this trial;
17. Any unstable condition or situation that may jeopardize patient safety and compliance;
18. Pregnancy or lactation in women of childbearing potential who have not taken adequate contraceptive measures;
19. Refusal to sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are pathological confirmed as rectal adenocarcinoma, clinical stage T3-4NxM0, and underwent the neoadjuvant therapy before surgical treatment.
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Area under curve(AUC) | through study completion, an average of 6 months
  Area under curve of prediction model

SECONDARY OUTCOMES:
Sensitivity | through study completion, an average of 6 months
  Sensitivity of prediction model
Specificity | through study completion, an average of 6 months
  Specificity of prediction model
Negative predictive value(NPV) | through study completion, an average of 6 months
  negative predictive value of prediction model
Positive predictive value(PPV) | through study completion, an average of 6 months
  positive predictive value of prediction model

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, Principal Investigator — Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yatsen University, Guangzhou, Guangdong, China